CLINICAL TRIAL: NCT03299322
Title: Clinical Assessment of Jia Wei Yang He Formula as a Plus Therapy in the Treatment of Persistent Asthma and Airway Microbiome Exploration Research
Brief Title: A Study to Assess Jia Wei Yang He Formula as a Plus Therapy in the Treatment of Persistent Asthma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Collaborators: Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2016LCSY098
Record Dates: First submitted 2017-09-21; First posted 2017-10-03 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2023-05

CONDITIONS: Bronchial Asthma
Keywords: Bronchial Asthma，TCM，microorganism
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: All treatment group received a standard anti-asthma treatment plus Jia Wei Yang He Formula on study entry, and the control group received Jia Wei Yang He Formula placebo instead.
Who Masked: Participant, Care Provider, Investigator
Masking Description: This is a Double-blind Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (Placebo Comparator): 80 participants will take oral therapy of 9.25 g Jia Wei Yang He granule Placebo twice a day for 28 consecutive days and also standard therapy of inhaled corticosteroid or beta2-agonist.
  Interventions: Drug: Jia Wei Yang He granule Placebo
- High dose Treatment Group (Experimental): Participants in high Jia Wei Yang He formula group will receive Jia Wei Yang He granule 18.5g twice a day for 28 consecutive days and also standard therapy of inhaled corticosteroid or beta2-agonist.
  Interventions: Drug: Jia Wei Yang He granule
- Low dose Treatment Group (Experimental): Participants in high Jia Wei Yang He formula group will receive Jia Wei Yang He granule 9.25g twice a day for 28 consecutive days and also standard therapy of inhaled corticosteroid or beta2-agonist.
  Interventions: Drug: Jia Wei Yang He granule

INTERVENTIONS:
Drug: Jia Wei Yang He granule — This is an empirical traditional Chinese medicine compound used in the treatment of asthma for a long time
  Other Names: Jia Wei Yang He Formula
  Arms: High dose Treatment Group; Low dose Treatment Group
Drug: Jia Wei Yang He granule Placebo — Made from 1/20 doses which has certain taste, but no therapeutic effect
  Other Names: Placebo
  Arms: Control Group

SUMMARY:
Investigators aimed to assess Jia Wei Yang He Formula as a plus therapy in the treatment of persistent asthma and to explore Airway Microbiome variation of Asthma by Traditional Chinese Medicine treatment

DETAILED DESCRIPTION:
Asthma is a common chronic inflammatory respiratory disease, patients showed high airway reactivity, and the clinical manifestations of recurrent wheezing, shortness of breath, chest tightness or cough with wheezing dyspnea mainly for a breath. Although many studies have shown that viral infections may be an important cause of asthma seasonal attacks. However, more and more studies have shown that bacterial infection is an important risk factor for asthma. Haemophilus influenzae, Moraxella Mora bacteria infection may increase the risk of asthma by a research report.

Chinese medicine decoction, as a common treatment for asthma, can significantly alleviate seasonal attacks and reduce the number of acute attacks. Research shows that Chinese medicine has widely immunomodulatory effects and imbalance of immune system in patients with asthma control, improve the cellular immunity of patients with airway and defense function, significantly reduced asthma attacks of which induced by upper airway infection or chronic persist asthma.

This study will be conducted for 4 weeks of standard anti-asthma treatment plus Jia Wei Yang He Formula for patients.Some patients are not willing to use standard treatment such as inhaled corticosteroids and long-acting β-adrenoceptor agonists because of side effects. We will provide these patients free JWYH formula after the efficacy of the JWYH is validated and the subsequent results are considered exploratory.

Participants will undergo a physical examination, lung function, blood and sputum collection and all induced sputum samples will be detected by 16S ribosomal RNA (16S rRNA) sequencing and analyzed for microbial bioinformatics. To study whether there is association between the efficacy of Jia Wei Yang He Formula and the changes in microbiota composition.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with chronic persistent asthma
* Annual uncontrollable time ≥ 3 months
* Patients who have given written informed consent

Exclusion Criteria:

* History of upper upper/lower respiratory infection in the previous 1 months
* History of long-term controller medication use for asthma (oral corticosteroid or intravenous corticosteroids therapy) within the preceding 1 months
* History of antibiotic use in the previous 1 months
* History of life-threatening asthma
* History of chronic lung diseases other than asthma, including but not limited to chronic obstructive pulmonary disease, bronchiectasis, emphysema, tuberculosis, sarcoidosis, pulmonary fibrosis, lung cancer, etc
* History of serious disease of the heart and cerebrovascular disease
* History of severe liver or renal dysfunction or disease
* History of severe disease in the hematopoietic system
* History of immunodeficiency (including, but not limited to, HIV positive detection, or other acquired or congenital immunodeficiency disease, or organ transplant history)
* History of any other condition (such as known drug or alcohol abuse or psychiatric disorder) which, in the opinion of the investigator, may preclude the patient from following and completing the protocol
* Are currently enrolled in, or discontinued within the last 30 days from, a clinical trial involving an investigational product or non-approved use of a drug or device (other than the investigational product used in this study), or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* History of allergies to the component of the investigated drugs
* Smoking within the past year
* Contraindication to induced sputum collection method on history or examination
* Any serious medical condition which, in the opinion of the Investigator, would pose a significant risk to the patient or interfere with the interpretation of safety, efficacy, or pharmacodynamic data

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Asthma Control Test Score variation | Baseline and 4 weeks
  Measured the change from Baseline to the end of treatment

SECONDARY OUTCOMES:
Airway microbial diversity | Baseline, 2 weeks and 4weeks
  Measured by 16S rRNA sequencing of induces sputum
Pulmonary function tests | Baseline and 4 weeks
  Measured the change from Baseline to the end of treatment
Fractional exhaled nitric oxide (FeNO) | Baseline and 4 weeks
  Measured the change from Baseline to the end of treatment of exhaled nitric oxide
Morning and evening Peak Expiratory Flow (PEF) | Measured during the 4 weeks treatment period
  Measured the change from Baseline to the end of treatment
Cytokine levels of serum | Baseline and 4 weeks
  Measured the change from Baseline to the end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Huiyong Zhang, Master, Study Chair — Longhua Hospital
Locations (8):
- China (8):
  - Longhua Hospital Affiliated Shanghai University of TCM, Shanghai, Shanghai Municipality
  - Fengxian District traditional Chinese medicine hospital, Shanghai
  - Jingan district center hospital, Shanghai
  - Pudong Hospital, Shanghai
  - Shanghai eighth people's hospital, Shanghai
  - Shanghai TCM-Integrated Hospital, Shanghai
  - Xuhui district center hospita, Shanghai
  - Zhongshan Hospital affiliated fudan university, Shanghai

REFERENCES:
- [Derived] Jiang W, Ma Z, Zhang H, Lynn HS, Xu B, Zhang X, Bi R, Fu J, Chen Y, Xiao Z, Zhang Z, Lu Z. Efficacy of Jia Wei Yang He formula as an adjunctive therapy for asthma: study protocol for a randomized, double blinded, controlled trial. Trials. 2018 Jul 4;19(1):355. doi: 10.1186/s13063-018-2739-8. PMID 29973284